CLINICAL TRIAL: NCT03290261
Title: Hypnosis as a Therapeutic Tool in Patients With Reccurent Cystitis
Acronym: HYPNOCYST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-PP-10
Record Dates: First submitted 2017-09-07; First posted 2017-09-21 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Reccurent Cystitis
MeSH Terms: interventions — Hypnosis

STUDY DESIGN:
Intervention Model Description: non-randomised, single center, pilote study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with reccurent cystitis (Experimental): Patient perform 3 hypnosis sessions
  Interventions: Other: Hypnosis

INTERVENTIONS:
Other: Hypnosis — 3 hypnosis sessions performed at 4 - 6 weeks apart

SUMMARY:
Half of the women present an episode of cystitis once in their lives. A recurrence occurs in about 20% to 30% of the patients, and half of these patients will make more than 4 episodes per year, defining recurrent cystitis (CR).

Complications such as pyelonephritis are rare (less than 0.5% of patients in the absence of underlying complication), however, CRs are responsible for a significant impact on women but also on society. Pain is at the forefront, but also the fear of not managing pollakiuria, with its social exclusion. The impact on sexuality is major. The medical circuit imposed on the patients is long and arduous. The clinical assessment sometimes reveals favorable factors, variable in pre- or post-menopause, but in the majority of cases, no explanatory cause can resolve the problem and some authors suggest resignation as a classic reaction to this problem. The only study on psychological disorders associated with recurrent cystitis suggests patients who are much more anxious than the average of female.

Hypnotherapy is an old technique, used for care in Western societies for at least two hundred years. By the word, the practitioner induces in the patient a particular state of consciousness characterized by an indifference on the outside and a hyper suggestibility. This "hypnotic" state of consciousness can be used to amplify the patient's internal resources to fight against anxiety and pain, and to eliminate symptoms.

The physiological mechanisms at work in hypnosis are the subject of recent studies becoming more and more precise. The results of these studies made it possible to objectify changes in cerebral functioning related to hypnotic trance.

A report by Inserm of 2015 confirms the effectiveness of this practice in hypnosedation, hypnoanalgesia and hypnotherapy, particularly in irritable bowel syndrome, although the methodology to be used in its evaluation is difficult and subjective. The principal investigator hypothesizes that the symptoms presented in recurrent cystitis (pain, anxiety) can be improved by hypnotherapy, and that thus the prognosis of this pathology can be totally modified.

In the absence of any study published in the literature, the investigator propose an intervention pilot study with minimal risks and constraints monocentric prospective non-randomized prospectively in 15 patients.

The main objective of this project is to demonstrate that hypnotherapy improves the psycho-emotional parameters of patients suffering from recurrent cystitis after 3 hypnosis sessions combined with home exercises performed by the patient. The evaluation will be carried out during the last session of hypnosis.

ELIGIBILITY:
Inclusion Criteria:

* Women aged at least 18 years
* Affiliated to social security
* Presenting recurrent cystitis defined by a frequency of more than 4 episodes per year, and alleging stress, pain, impaired quality of life or anxiety related to this condition.
* Available to perform 3 hypnosis sessions of one hour to 4/6 weeks apart and to perform home task prescriptions (self-hypnosis or hearing of a recorded medium).
* Having previously been explored according to good practice and informed with the tool created by the RéSO InfectiO PACA Est, with a 3 months follow-up compared to this initial consultation.
* Having signed informed consent.
* Patient under tutelage, under curatorship, protected by the law

Exclusion Criteria:

* Pregnant women (declarative because no theoretical contraindication, but different care)
* Other nonpharmacological treatments (acupuncture, cognitive and behavioral therapy, sophrology ...)
* Treatment with psychotropic drugs modified for less than six months
* Severe visceral deficiencies in the previous year.
* Individual psychiatric pathology
* Other progressive infectious diseases requiring antibiotic treatments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2020-10-29 (Actual)

PRIMARY OUTCOMES:
Score at HAD Scale | Month 3
  Overall score at the HAD scale at the end of treatment ie M3, compared to the initial score.

SECONDARY OUTCOMES:
Score at Pain evaluation scale | Month 3
  Overall score at the Pain evaluation scale at the end of treatment ie M3, compared to the initial score.
Evolution of HAD scale score | Month 12
Evolution of Pain evaluation scale score | Month 12
Patient satisfaction | Month 12
  Patient satisfaction will be assessed on a simple numerical scale of 1 to 10 at the end of treatment
Ability to manage the symptoms | Month 12
  The ability to manage their symptoms sera evaluated by a semantic scale at the end of treatment
Sexuality evaluation | Month 12
  Assessment of the performance in charge of sexuality serum evaluation of the overall semantic scale and on the specific improvement of 2 criteria: anxiety of the sexual act, comfort (dyspareunia) during the act.
Consumption of heath care | Month 12
  Consumption of health care compared to the previous year (medical consultations for cystitis, number of laboratory tests, antibiotics or analgesics, work stoppage)

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Mondain, PH, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Hôpital Archet, Nice, France